CLINICAL TRIAL: NCT04210193
Title: Is Intralymphatic Allergen Immunotherapy Effective and Safe: a Human Randomized Clinical Trial- Substudy Borås With a Randomized Preseasonal Booster
Brief Title: Is Intralymphatic Allergen Immunotherapy Effective and Safe?
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lars Olaf Cardell (Other)
Responsible Party: Sponsor-Investigator, Lars Olaf Cardell, Professor, Karolinska Institutet
Organization: Karolinska Institutet (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ILIT Borås EPN 2014/251
Record Dates: First submitted 2019-12-17; First posted 2019-12-24 (Actual); Last update posted 2019-12-24 (Actual); Status verified 2019-12

CONDITIONS: Allergic Rhinitis Due to Grass Pollen
MeSH Terms: interventions — Serum Albumin, Human

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active booster (Active Comparator): After three basic open label grass allergen ILIT injections the patient is randomized to an active ILIT booster 1 year after the first treatment.
  Interventions: Drug: ALK Alutard 5-grasses
- Placebo booster (Placebo Comparator): After three basic open label grass allergen ILIT injections the patient is randomized to a placebo ILIT booster 1 year after the first treatment.
  Interventions: Drug: ALK Diluent

INTERVENTIONS:
Drug: ALK Alutard 5-grasses — 0.1 mL of 10 000 SQ-U/mL (1000 SQ-U) as an intralymphatic injection
  Other Names: Grass allergen with aluminum adjuvant
  Arms: Active booster
Drug: ALK Diluent — 0.1 mL of ALK Diluent as an intralymphatic injection
  Other Names: Human albumin
  Arms: Placebo booster

SUMMARY:
15 patients with moderate to severe allergic rhinitis against grass were recruited and enrolled in the study. They received three open label intralympatic grass allergen injections with the dose 1000 SQ-U each and with one month interval. The next year the patients were randomized double blind to an active or placebo booster injection of 1000 SQ-U before the pollen season. Grass specific IgG4 levels were measured before and at various time ponts after treatment.

DETAILED DESCRIPTION:
The purpose of the study is to evaluate whether intralymphatic administration of AIT is a safe and effective treatment for patients with pollen-induced allergic rhinitis. The long term goal is to provide a base for a more efficient administration of ASIT, which will reduce both the dose necessary and the number of clinic visits associated with the conventional subcutaneous ASIT.

The aim of the present substudy is to evaluate if a randomized preseasonal ILIT booster, after three open label ILIT injections, can increase the allergen specific IgG4 antibodies, and if the IgG4 increase can be correlated to clinical effect characterized with seasonal questionnaires.

The first part of the study is completed and published (PMID: 23374268)

ELIGIBILITY:
Inclusion Criteria:

* Age 18-50,
* Seasonal allergic symptoms for birch and/or grass verified by skin prick test,
* Accepted informed consent

Exclusion Criteria:

* Pregnancy or nursing
* Autoimmune or collagen disease (known)
* Cardiovascular disease
* Perennial pulmonary disease
* Hepatic disease
* Renal disease
* Cancer
* Any medication with a possible side-effect of interfering with the immune response
* Previous immuno- or chemotherapy
* Chronic diseases
* Other upper airway disease (non-allergic sinusitis, nasal polyps, chronic obstructive and restrictive lung disease)
* Disease or conditions rendering the treatment of anaphylactic reactions difficult (symptomatic coronary heart diseases, severe arterial hypertension and treatment with β-blockers)
* Major metabolic disease
* Known or suspected allergy to the study product
* Alcohol or drug abuse
* Mental incapability of coping with the study
* Withdrawal of informed consent

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2014-04-25 (Actual); Primary Completion 2019-12-01 (Actual); Study Completion 2019-12-01 (Actual)

PRIMARY OUTCOMES:
Change in the serum-level of timothy specific IgG4 after 1 month | Change between baseline and 1 month after treatment.
  Blood samples with measurement of allergen specific blocking IgG4 antibodies
Change in the serum-level of timothy specific IgG4 after 9 months | Change between baseline and 9 months after treatment.
  Blood samples with measurement of allergen specific blocking IgG4 antibodies
Change in the serum-level of timothy specific IgG4 2 months after booster | Change between baseline and 2 months after the booster treatment (14 months after the basic treatment).
  Blood samples with measurement of allergen specific blocking IgG4 antibodies
Change in the serum-level of timothy specific IgG4 10 months after booster | Change between baseline and 10 months after the booster treatment (22 months after the basic treatment).
  Blood samples with measurement of allergen specific blocking IgG4 antibodies

CONTACTS AND LOCATIONS:
Overall Officials: Lars Olaf Cardell, Professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Allergy Unit, Södra Älvsborgs Hospital, Borås, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hylander T, Larsson O, Petersson-Westin U, Eriksson M, Kumlien Georen S, Winqvist O, Cardell LO. Intralymphatic immunotherapy of pollen-induced rhinoconjunctivitis: a double-blind placebo-controlled trial. Respir Res. 2016 Jan 27;17:10. doi: 10.1186/s12931-016-0324-9. PMID 26817454
- [Background] Konradsen JR, Grundstrom J, Hellkvist L, Tran TAT, Andersson N, Gafvelin G, Kiewiet MBG, Hamsten C, Tang J, Parkin RV, Shamji MH, Hedlin G, Cardell LO, van Hage M. Intralymphatic immunotherapy in pollen-allergic young adults with rhinoconjunctivitis and mild asthma: A randomized trial. J Allergy Clin Immunol. 2020 Mar;145(3):1005-1007.e7. doi: 10.1016/j.jaci.2019.11.017. Epub 2019 Nov 24. No abstract available. PMID 31775016
- [Derived] Weinfeld D, Westin U, Hellkvist L, Mellqvist UH, Jacobsson I, Cardell LO. A preseason booster prolongs the increase of allergen specific IgG4 levels, after basic allergen intralymphatic immunotherapy, against grass pollen seasonal allergy. Allergy Asthma Clin Immunol. 2020 Apr 28;16:31. doi: 10.1186/s13223-020-00427-z. eCollection 2020. PMID 32368217